CLINICAL TRIAL: NCT00686556
Title: Total Marrow Irradiation and Myeloablative Chemotherapy Followed By Double Umbilical Cord BloodTransplantation In Patients With Refractory Acute Leukemia
Brief Title: Total Marrow Irradiation for Refractory Acute Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007LS024; MT2006-24 (Other: Blood and Marrow Transplantation Program); 0708M14041 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-05-29; First posted 2008-05-30 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome; Multiple Myeloma
Keywords: recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); ALL; MDS
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Multiple Myeloma; Leukemia, Myeloid, Acute; Congenital Abnormalities | interventions — Cyclophosphamide; Cyclosporine; fludarabine; fludarabine phosphate; Mycophenolic Acid; Cord Blood Stem Cell Transplantation; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort -1 (Experimental): Patient receives preparative therapy including Fludarabine, cyclophosphamide, and total marrow irradiation of 12 Gy on Days -4 through -1, and starts immunosuppressive therapy using cyclosporine, Mycophenolate Mofetil, followed by umbilical cord blood transplantation, or HLA-matched related donor bone marrow transplantation and granulocyte colony-stimulating factor administration.
  Interventions: Drug: cyclophosphamide; Drug: cyclosporine; Drug: Fludarabine; Drug: mycophenolate mofetil; Radiation: total marrow irradiation; Procedure: umbilical cord blood transplantation; Biological: Granulocyte colony-stimulating factor; Biological: HLA-matched related donor bone marrow
- Cohort 1 (Experimental): Patient receives preparative therapy including Fludarabine, cyclophosphamide, and total marrow irradiation of 15 Gy on Days -5 through -1, and starts immunosuppressive therapy using cyclosporine, Mycophenolate Mofetil, followed by umbilical cord blood transplantation, or HLA-matched related donor bone marrow transplantation and granulocyte colony-stimulating factor administration.
  Interventions: Drug: cyclophosphamide; Drug: cyclosporine; Drug: Fludarabine; Drug: mycophenolate mofetil; Radiation: total marrow irradiation; Procedure: umbilical cord blood transplantation; Biological: Granulocyte colony-stimulating factor; Biological: HLA-matched related donor bone marrow
- Cohort 2 (Experimental): Patient receives preparative therapy including Fludarabine, cyclophosphamide, and total marrow irradiation of 18 Gy on Days -6 through -1, and starts immunosuppressive therapy using cyclosporine, Mycophenolate Mofetil, followed by umbilical cord blood transplantation, or HLA-matched related donor bone marrow transplantation and granulocyte colony-stimulating factor administration.
  Interventions: Drug: cyclophosphamide; Drug: cyclosporine; Drug: Fludarabine; Drug: mycophenolate mofetil; Radiation: total marrow irradiation; Procedure: umbilical cord blood transplantation; Biological: Granulocyte colony-stimulating factor; Biological: HLA-matched related donor bone marrow
- Cohort 3 (Experimental): Patient receives preparative therapy including Fludarabine, cyclophosphamide, and total marrow irradiation of 21 Gy on Days -7 through -1, and starts immunosuppressive therapy using cyclosporine, Mycophenolate Mofetil, followed by umbilical cord blood transplantation, or HLA-matched related donor bone marrow transplantation and granulocyte colony-stimulating factor administration.
  Interventions: Drug: cyclophosphamide; Drug: cyclosporine; Drug: Fludarabine; Drug: mycophenolate mofetil; Radiation: total marrow irradiation; Procedure: umbilical cord blood transplantation; Biological: Granulocyte colony-stimulating factor; Biological: HLA-matched related donor bone marrow
- Cohort 4 (Experimental): Patient receives preparative therapy including Fludarabine, cyclophosphamide, and total marrow irradiation of 24 Gy on Days -8 through -1, and starts immunosuppressive therapy using cyclosporine, Mycophenolate Mofetil, followed by umbilical cord blood transplantation, or HLA-matched related donor bone marrow transplantation and granulocyte colony-stimulating factor administration.
  Interventions: Drug: cyclophosphamide; Drug: cyclosporine; Drug: Fludarabine; Drug: mycophenolate mofetil; Radiation: total marrow irradiation; Procedure: umbilical cord blood transplantation; Biological: Granulocyte colony-stimulating factor; Biological: HLA-matched related donor bone marrow

INTERVENTIONS:
Drug: cyclophosphamide — 60 mg/kg/day intravenous x 2 days pre-transplant, total dose 120 mg/kg
  Other Names: Cytoxan
Drug: cyclosporine — Beginning on Day -3 pre-transplant maintaining a level of >200 ng/mL. CSA dosing will be monitored and altered as clinically appropriate by Pharm D or physician, and discontinue at approximately day + 180 post-transplant.
  Other Names: CSA
Drug: Fludarabine — 25 mg/m2/day intravenous as a 1 hour infusion for consecutive 3 days pre-transplant, total dose 75 mg/m2
  Other Names: Fludara
Drug: mycophenolate mofetil — Beginning on day -3, use intravenous route between days -3 and +5, followed by oral administration on Day +6 through +30, if tolerated. 15mg/kg/dose for patients <40 kg, 3 gm/day for patients >40 kg.
  Other Names: MMF
Radiation: total marrow irradiation — Dose escalating schedule per Cohort (TMI: 300 cGy) once daily.
  Other Names: TMI
Procedure: umbilical cord blood transplantation — product will be infused via intravenous drip on Day 0 according to current University of Minnesota guidelines for Umbilical Cord Blood Grafts
  Other Names: umbilical cord blood; allogeneic hematopoietic stem cell transplantation
Biological: Granulocyte colony-stimulating factor — 5 mcg/kg/day intravenous or subcutaneous based on body weight beginning on Day +1 after umbilical cord blood infusion until absolute neutrophil count exceeds 2.5 x 10^9/L for 3 consecutive days.
  Other Names: G-CSF
Biological: HLA-matched related donor bone marrow — Related donor bone marrow or mobilized stem cells will be collected (target cell dose 5x10^8 nucleated cells/kg recipient weight, minimum 3x10^8 nucleated cells/kg recipient weight) and infused without processing on day 0 according to University of Minnesota Blood and Marrow Transplant Program guidelines.
  Other Names: mobilized peripheral blood stem cells

SUMMARY:
RATIONALE: Giving chemotherapy and total marrow irradiation before a donor umbilical cord blood or hematopoietic stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening.

PURPOSE: This phase I trial is studying the side effects and best dose of total marrow irradiation when given together with combination chemotherapy and umbilical cord blood hematopoietic stem cell transplant in treating patients with acute leukemia, acute myeloid leukemia or multiple myeloma that did not respond to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of total marrow irradiation (TMI) delivered by image-guided tomographic intensity-modulated radiotherapy when administered in combination with myeloablative chemotherapy in patients undergoing double umbilical cord blood (UCB) transplantation or hematopoietic stem cell for refractory acute leukemia.

Secondary

* Determine the incidence of engraftment (defined as achievement of neutrophil count > 500/uL at 42 days after transplantation).
* Determine the incidence of platelet engraftment at 6 months and at 1 year after transplantation.
* Evaluate the incidence of complete donor chimerism and the relative contribution of each UCB unit to donor engraftment within the first 100 days after transplantation.
* Determine the incidence of transplantation-related mortality (TRM) at 6 months after treatment with a TMI-containing myeloablative conditioning regimen.
* Determine the incidence of grade II-IV and grade III-IV acute graft-versus-host disease (GVHD) at 100 days after transplantation.
* Determine the incidence of chronic GVHD at 1 year after transplantation.
* Determine the incidence of relapse at 1 year after transplantation.
* Determine the survival and disease-free survival at 1 and 2 years after transplantation.
* Assess the durability of remission based on presence of rapid early response (defined by clearance of leukemic blasts from the bone marrow at 21 days after transplantation).

OUTLINE: This is a dose-escalation study of total marrow irradiation (TMI).

* Myeloablative conditioning regimen: Patients receive fludarabine phosphate IV over 1 hour once daily for 3 days between days -12 and -6 and cyclophosphamide IV once daily for 2 days between days -11 and -6. Patients undergo TMI once daily for 4-8 days between days -8 and -1.
* Donor umbilical cord blood (UCB) transplantation: Patients undergo single-unit or double-unit donor UCB transplantation on day 0. Patients receive filgrastim (G-CSF) IV or subcutaneously once daily beginning on day 1 and continuing until blood counts recover.
* Related Donor: Related donor bone marrow will be collected (target cell dose 5x10^8 nucleated cells/kg recipient weight, minimum 3x10^8 nucleated cells/kg recipient weight) and infused without processing on day 0.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive cyclosporine IV over 2 hours or orally 2-3 times daily beginning on day -3 and continuing until day 100, followed by a taper until day 180, in the absence of GVHD. Patients also receive mycophenolate mofetil IV or orally 2-3 times daily beginning on day -3 and continuing until day 30 (or 7 days after engraftment), in the absence of acute GVHD.

Patients are followed periodically for up to 2 years after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia

  * ≥ Complete remission 2 (CR2) (adults ≥ 18 years and ≤ 55 years)
  * CR2 in pediatrics (defined as <18 years) and <12 months duration of first remission
  * ≥ CR3 or not in remission (pediatric patients <18 years)
  * T cell leukemia ≥ CR2
  * Evidence of pre-transplant minimal residual disease (MRD) by flow cytometry, FISH or cytogenetics
* Myelodysplastic syndrome

  * ≤ 55 years of age and ≥ 10% blasts, not responsive to hypomethylating agents and/or conventional therapy
* Acute myeloid leukemia

  * Not in remission (pediatric patients <18 years)
  * Not in remission (10-30% blasts in the bone marrow for adult patients ≥18 years and ≤ 55 years)
  * Evidence of pre-transplant minimal residual disease (MRD) by flow cytometry, FISH or cytogenetics
* Multiple myeloma

  * No prior autologous transplant and fitting into one of the following disease categories:

    * Early disease stage (CR1/PR1) with high-risk molecular features
    * Early disease stage (CR1/PR1) with high-risk clinical features
    * Late disease stage (CR2/PR2+) with high-risk clinical features
* Other high risk hematologic malignancies - to be approved by 2 or more hematology/oncology and BMT physicians
* Patients with prior CNS involvement are eligible provided that it has been treated and is in remission. CNS therapy (chemotherapy or radiation) should continue as medically indicated during the protocol.
* Have acceptable organ function within 14 days of study registration defined as:

  * Renal: glomerular filtration rate > 60ml/min/1.73m2
  * Hepatic: bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), Alkaline phosphatase (ALP) < 5 x upper limit of normal (ULN)
  * Pulmonary function: Carbon Monoxide Diffusing Capacity corrected (DLCOcorr) > 50% of normal, (oxygen saturation [>92%] can be used in child where pulmonary function tests (PFT's) cannot be obtained)
  * Cardiac: left ventricular ejection fraction ≥ 45% by echocardiogram (ECHO) or multi gated acquisition scan (MUGA)
* Karnofsky performance status (PS) >80% for ages 16 years and older or Lansky Play Score >50 for < 16 years
* An acceptable source of stem cells according to current University of Minnesota BMT program guidelines:

  * UCB graft will be composed of two partially HLA matched units. Each unit must be matched at 4-6 HLA loci to the recipient and to each other. If two matched units are not available, then a single HLA 4-6 matched unit may be used if of adequate cell dose - total graft dose must be >3 x 107 MNC/kg
  * HLA-matched related donor (6/6 or 5/6 antigen match)
  * HLA-matched unrelated adult donor (if previously identified)
* Women of childbearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment.
* Voluntary written consent

Exclusion Criteria:

* Active uncontrolled infection at time of enrollment or documented fungal infection within 3 months.
* Evidence of Human immunodeficiency virus (HIV) infection
* Pregnant or breast feeding. The agents used in this study may be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy.
* Prior myeloablative transplant within the last 6 months
* Prior total body irradiation (TBI) making total marrow irradiation (TMI) not feasible

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of total marrow irradiation (TMI) | Day 42 and 6 months
  Maximum tolerated dose (MTD) is the highest dose of a drug or treatment that does not cause unacceptable side effects. The MTD of TMI will be determined by using the modified Continual Reassessment Method (CRM). The goal of this CRM will be to identify 1 of the 5 dose levels which corresponds to the desired maximum toxicity rate of <=15%.

SECONDARY OUTCOMES:
Incidence of neutrophil engraftment | Day 42
  Neutrophil engraftment is defined as the first day of three consecutive days where the neutrophil count (absolute neutrophil count) is 500 cells/mm3 (0.5 x 109/L) or greater.
Incidence of platelet engraftment | 6 Months and 1 Year After Transplantation
  Platelet engraftment is defined as 20,000/mm^3 (20 x 10^9/L) for 3 consecutive days unsupported by a platelet transfusion.
Incidence of complete donor chimerism | Day 100
  Defined as a state in bone marrow transplantation in which bone marrow and host cells exist compatibly without signs of graft-versus-host rejection disease.
Incidence of transplantation-related mortality | 6 Months
  In the field of transplantation, toxicity is high and all deaths without previous relapse or progression are usually considered as related to transplantation.
Incidence of grade II-IV and grade III-IV acute graft-versus-host disease (GVHD) after transplantation | Day 100
  Acute Graft-Versus-Host Disease is a severe short-term complication created by infusion of donor cells into a foreign host.
Incidence of chronic GVHD after transplantation | 1 Year
  Chronic Graft-Versus-Host Disease is a severe long-term complication created by infusion of donor cells into a foreign host.
Incidence of relapse after transplantation | 1 Year
  The return of disease after its apparent recovery/cessation.
Disease-free survival after transplantation | 1 year and 2 years
  Disease-free survival (progression-free survival [PFS]) is the length of time during and after medication or treatment during which the disease being treated (usually cancer) does not get worse. It is sometimes used as a metric to study the health of a person with a disease to try to determine how well a new treatment is working.
Durability of remission based on presence of rapid early response after transplantation | Day 21
  Remission - a decrease in or disappearance of signs and symptoms of cancer. In partial remission, some, but not all, signs and symptoms of cancer have disappeared. In complete remission, all signs and symptoms of cancer that can be detected with modern technology have disappeared, although cancer still may be in the body.
Overall survival after transplantation | 1 year and 2 years
  The percentage of people in a study or treatment group who are alive for a certain period of time after they were diagnosed with or treated for a disease, such as cancer.

CONTACTS AND LOCATIONS:
Overall Officials: John Wagner, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States